CLINICAL TRIAL: NCT04677387
Title: Addressing the Opioid Epidemic Through Community Pharmacy Engagement: Randomized Controlled Trial (Aim 2)
Brief Title: Nalox-Comm: Naloxone Communication Training for Pharmacists
Acronym: Nalox-Comm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 20-2192; R34DA046598 (NIH)
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2023-10

CONDITIONS: Naloxone
Keywords: community pharmacy; communication
MeSH Terms: conditions — Communication | interventions — Pharmacists

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prescribe to Prevent Naloxone Training Module (Placebo Comparator): This a 55-minute online module that covers basic information about naloxone that is relevant to community pharmacists.
  Interventions: Behavioral: Prescribe to Prevent: Overdose Prevention and Naloxone Rescue Kits for Prescribers and Pharmacists
- Nalox-Comm (Experimental): This is a newly developed 30-60 minute online module focused on teaching pharmacists how to overcome naloxone communication barriers.
  Interventions: Behavioral: Nalox-comm Training Module

INTERVENTIONS:
Behavioral: Nalox-comm Training Module — The online communication module will be 30-60 minutes. Content will include: 1) using non-judgmental language, 2) how to raise the topic of overdose (OD) and naloxone with patients in a non-threatening manner; 3) videos modeling how to initiate the conversation with patients and caregivers; 4) considerations in how to communicate differently with patients versus caregivers; and 5) addressing pharmacists' perceived barriers to naloxone counseling. Pharmacists can receive continuing education credit (0.1 CEU) for completing the course.
  Arms: Nalox-Comm
Behavioral: Prescribe to Prevent: Overdose Prevention and Naloxone Rescue Kits for Prescribers and Pharmacists — A 55 minute long online module with videos, didactic content, and quizzes that covers the following topics: risk factors for overdose (OD), how to respond to OD, how naloxone works, types of naloxone, how to administer naloxone, medico-legal issues, how to bill for naloxone, and strategies to address overdose. Pharmacists can receive continuing education credit (0.125 CEUs) for completing the course.
  Arms: Prescribe to Prevent Naloxone Training Module

SUMMARY:
This is a pilot Randomized Controlled Trial (RCT) in which 120 pharmacists will be randomized to an experimental or control group and data on naloxone dispensing and secondary outcomes will be collected over the course of the RCT.

DETAILED DESCRIPTION:
This is a prospective pilot RCT that will evaluate the impact of naloxone communication training (Nalox-Comm) on 120 pharmacists' naloxone dispensing behaviors (primary outcome). Data will be collected at baseline, immediately after training is completed, and at 3-month follow up. Data sources include pharmacy records (for naloxone dispensing), simulated patient observations (to rate quality of communication), and survey data (for self-reports of knowledge and self-efficacy).

ELIGIBILITY:
Inclusion Criteria:

* currently work at a pharmacy that stocks naloxone;
* currently work at a rural community pharmacy;
* are at least 18 years of age; and
* speak English.

Exclusion Criteria:

* Non-staff pharmacists such as pharmacy "floaters" or fill-in pharmacists will not be eligible to participate.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Delesha Carpenter, PhD, MSPH, Principal Investigator — UNC Eshelman School of Pharmacy
Locations (1):
- University of North Carolina at Chapel Hill (Asheville campus), Asheville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: SAP, ICF
Time Frame: 9-36 months following publication
Access Criteria: The investigator who proposes to use the data must have IRB, IEC, or REB approval, as applicable, and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Thornton JD, Lyvers E, Scott VGG, Dwibedi N. Pharmacists' readiness to provide naloxone in community pharmacies in West Virginia. J Am Pharm Assoc (2003). 2017 Mar-Apr;57(2S):S12-S18.e4. doi: 10.1016/j.japh.2016.12.070. Epub 2017 Feb 2. PMID 28163027
- [Background] Hagemeier NE, Murawski MM, Lopez NC, Alamian A, Pack RP. Theoretical exploration of Tennessee community pharmacists' perceptions regarding opioid pain reliever abuse communication. Res Social Adm Pharm. 2014 May-Jun;10(3):562-75. doi: 10.1016/j.sapharm.2013.07.004. Epub 2013 Aug 24. PMID 23981913
- [Background] Gamm L, Stone S, Pittman S. Mental health and mental disorders-A rural challenge: A literature review. Rural healthy people. 2010;1:97-114.
- [Background] Browne T, Priester MA, Clone S, Iachini A, DeHart D, Hock R. Barriers and Facilitators to Substance Use Treatment in the Rural South: A Qualitative Study. J Rural Health. 2016 Winter;32(1):92-101. doi: 10.1111/jrh.12129. Epub 2015 Jul 15. PMID 26184098
- [Background] Freeman PR, Goodin A, Troske S, Strahl A, Fallin A, Green TC. Pharmacists' role in opioid overdose: Kentucky pharmacists' willingness to participate in naloxone dispensing. J Am Pharm Assoc (2003). 2017 Mar-Apr;57(2S):S28-S33. doi: 10.1016/j.japh.2016.12.064. Epub 2017 Jan 28. PMID 28139459
- [Background] Mueller SR, Koester S, Glanz JM, Gardner EM, Binswanger IA. Attitudes Toward Naloxone Prescribing in Clinical Settings: A Qualitative Study of Patients Prescribed High Dose Opioids for Chronic Non-Cancer Pain. J Gen Intern Med. 2017 Mar;32(3):277-283. doi: 10.1007/s11606-016-3895-8. Epub 2016 Oct 31. PMID 27798775
- [Background] Nielsen S, Menon N, Larney S, Farrell M, Degenhardt L. Community pharmacist knowledge, attitudes and confidence regarding naloxone for overdose reversal. Addiction. 2016 Dec;111(12):2177-2186. doi: 10.1111/add.13517. Epub 2016 Aug 16. PMID 27367125
- [Background] Liekens S, Vandael E, Roter D, Larson S, Smits T, Laekeman G, Foulon V. Impact of training on pharmacists' counseling of patients starting antidepressant therapy. Patient Educ Couns. 2014 Jan;94(1):110-5. doi: 10.1016/j.pec.2013.09.023. Epub 2013 Oct 12. PMID 24169022
- [Background] Alte D, Weitschies W, Ritter CA. Evaluation of consultation in community pharmacies with mystery shoppers. Ann Pharmacother. 2007 Jun;41(6):1023-30. doi: 10.1345/aph.1H565. Epub 2007 May 22. PMID 17519295
- [Background] Weiss MC, Booth A, Jones B, Ramjeet S, Wong E. Use of simulated patients to assess the clinical and communication skills of community pharmacists. Pharm World Sci. 2010 Jun;32(3):353-61. doi: 10.1007/s11096-010-9375-z. Epub 2010 Mar 18. PMID 20238164
- [Background] Madden JM, Quick JD, Ross-Degnan D, Kafle KK. Undercover careseekers: simulated clients in the study of health provider behavior in developing countries. Soc Sci Med. 1997 Nov;45(10):1465-82. doi: 10.1016/s0277-9536(97)00076-2. PMID 9351137
- [Background] Bjornsdottir I, Granas AG, Bradley A, Norris P. A systematic review of the use of simulated patient methodology in pharmacy practice research from 2006 to 2016. Int J Pharm Pract. 2020 Feb;28(1):13-25. doi: 10.1111/ijpp.12570. Epub 2019 Aug 9. PMID 31397533
- [Background] Wilson JD, Spicyn N, Matson P, Alvanzo A, Feldman L. Internal medicine resident knowledge, attitudes, and barriers to naloxone prescription in hospital and clinic settings. Subst Abus. 2016 Jul-Sep;37(3):480-487. doi: 10.1080/08897077.2016.1142921. Epub 2016 Jan 28. PMID 26820604
- [Background] Williams AV, Strang J, Marsden J. Development of Opioid Overdose Knowledge (OOKS) and Attitudes (OOAS) Scales for take-home naloxone training evaluation. Drug Alcohol Depend. 2013 Sep 1;132(1-2):383-6. doi: 10.1016/j.drugalcdep.2013.02.007. Epub 2013 Feb 28. PMID 23453260
- [Background] Strahan R, Gerbasi K. Short, homogenous version of the Marlowe-Crowne social desirability scale. Journal of Clinical Psychology. 1972;28(191):193.
- [Background] Diggle P, Heagerty P, Liang K-Y, Zeger S. Analysis of longitudinal data. Oxford University Press; 2002.
- See also: Parker T. Rural-Urban Continuum Codes. 2013. — https://www.ers.usda.gov/data-products/rural-urban-continuum-codes.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Prescribe to Prevent Naloxone Training Module: This is a 55-minute online module that covers basic information about naloxone that is relevant to community pharmacists.
  Prescribe to Prevent: Overdose Prevention and Naloxone Rescue Kits for Prescribers and Pharmacists: A 55 minute long online module with videos, didactic content, and quizzes that covers the following topics: risk factors for overdose (OD), how to respond to OD, how naloxone works, types of naloxone, how to administer naloxone, medico-legal issues, how to bill for naloxone, and strategies to address overdose. Pharmacists can receive continuing education credit (0.125 CEUs) for completing the course.
Period: Overall Study
Arm/Group | Prescribe to Prevent Naloxone Training Module | Nalox-Comm
Started | 25 | 23
Baseline Survey | 25 | 23
Immediate Post-training Survey | 18 | 19
1-month Follow-up Simulated Patient Data | 17 | 16
3-month Follow-up Survey | 17 | 18
3-month Follow-up Dispensing Data | 19 | 20
Completed | 17 | 18
Not Completed | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prescribe to Prevent Naloxone Training Module | Nalox-Comm | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 22 | 46
  >=65 years | 1 | 1 | 2
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender: Female | 16 | 11 | 27
  Sex/Gender: Male | 8 | 12 | 20
  Sex/Gender: Prefer not to answer | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 24 | 23 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 22 | 21 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 23 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change in Naloxone Dispensing Rate Over a 6-month Period
Description: Pharmacy records indicated the number of times each pharmacy dispensed naloxone and opioid prescriptions over the RCT period. These data were aggregated into the total number of naloxone and opioid prescriptions dispensed in the 3 months pre-intervention and the 3 months post-intervention.
  The change in naloxone dispensing rates was measured by comparing pharmacy records of the number of naloxone products dispensed in the three months prior to study participation to the number of naloxone products dispensed in the three months after study completion. The rate was defined as the number of naloxone products dispensed divided by the number of opioid prescriptions dispensed in each 3-month period.
Time Frame: 3-month period before intervention and 3-month follow-up dispensing data
Measure: Mean (Standard Deviation); unit: number of naloxone products dispensed
Arm/Group | Prescribe to Prevent Naloxone Training Module | Nalox-Comm
Number analyzed (Participants) | 19 | 20
number of naloxone products dispensed | .0073 (.015) | .0041 (.0139)
Statistical Analysis 1: Comparison: Prescribe to Prevent Naloxone Training Module vs Nalox-Comm; Test type: Superiority; p = 0.473, Regression, Linear; Linear regression using a Generalized Estimating Equation (GEE) model clustering on pharmacy; Mean Difference (Final Values) = -.00325

2. Secondary Outcome: Mean Willingness to Dispense Naloxone Score
Description: An online survey including 6 self-reported Likert-scale items will assess pharmacists' willingness to dispense naloxone. These items assess pharmacists' willingness to engage in naloxone counseling activities, including educating patients to recognize overdose and administer naloxone, proactively identify individuals for naloxone dispensation and dispense naloxone. Response options will range from 1= "not at all willing" to 4= "very willing." Items were averaged to create a mean willingness score (range = 1-4), with higher scores indicating more willingness to dispense naloxone.
Time Frame: up to 3-month Follow-up Survey
Population: Only participants who completed Baseline and 3-month Follow-up Survey were analyzed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Prescribe to Prevent Naloxone Training Module | Nalox-Comm
Number analyzed (Participants) | 17 | 18
score on a scale
  Baseline Survey | 3.72 (0.07) | 3.57 (0.117)
  Immediate Post-training Survey | 3.64 (0.096) | 3.84 (0.07)
  3-month Follow-up Survey | 3.47 (0.14) | 3.69 (0.107)
Statistical Analysis 1: Comparison: Prescribe to Prevent Naloxone Training Module vs Nalox-Comm; Test type: Superiority; p = .007, Regression, Linear; Linear regression with Generalized Estimating Equation (GEE) model

3. Secondary Outcome: Mean Naloxone Counselling Self-Efficacy Score
Description: An online survey including 6 self-reported Likert-scale items assessed pharmacists' self-efficacy to counsel about naloxone. Pharmacists rated their confidence to engage in various naloxone communication tasks including: engage in naloxone counseling when the pharmacy is busy and discuss naloxone in a way that does not offend customers. Response options ranged from 1= "not at all confident" to 4= "very confident." Items were averaged to create a mean self-efficacy score (range = 1-4), with higher scores indicating greater self-efficacy to dispense naloxone.
Time Frame: up to 3-month Follow-up Survey
Population: Only participants who completed Baseline and 3-month Follow-up Survey were analyzed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Prescribe to Prevent Naloxone Training Module | Nalox-Comm
Number analyzed (Participants) | 17 | 18
score on a scale
  Baseline Survey | 3.08 (.012) | 2.74 (0.112)
  Immediate Post-training Survey | 3.19 (0.116) | 3.4 (0.107)
  3-month Follow-up Survey | 3.28 (0.105) | 3.51 (0.098)
Statistical Analysis 1: Comparison: Prescribe to Prevent Naloxone Training Module vs Nalox-Comm; Test type: Superiority; p = .002, Regression, Linear; Linear regression with a Generalized Estimating Equation (GEE) model

4. Secondary Outcome: Mean Pharmacist Quality of Non-verbal Communication Score
Description: Simulated patients (SPs) called pharmacists and used a validated observation guide that has been adapted for use for telephone interactions to rate the pharmacists' quality of non-verbal communication. The guide included 4 items (i.e., explained things clearly, listened carefully, showed respect, and spent enough time with the SP) measured on a 5-point scale (1= not at all satisfied, 2= partly satisfied, 3= satisfied, 4= more than satisfied, 5= very satisfied). Higher scores (range = 1-5) indicate a more positive evaluation of the interaction.
Time Frame: up to 1-month post-training
Population: All available data are reported and include pharmacists whose communication behavior was possible to be observed.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Prescribe to Prevent Naloxone Training Module | Nalox-Comm
Number analyzed (Participants) | 17 | 16
score on a scale
  baseline | 3.31 (0.141) | 3.5 (0.149)
  1-month follow-up | 3.62 (0.182) | 4.11 (0.123)
Statistical Analysis 1: Comparison: Prescribe to Prevent Naloxone Training Module vs Nalox-Comm; Test type: Superiority; p = 0.169, Regression, Linear; Linear regression with Generalized Estimating Equation (GEE) model

ADVERSE EVENTS:
Time Frame: From the time of informed consent provision through 3-month follow-up survey, a total of up to 6 months.
Arm/Group | Prescribe to Prevent Naloxone Training Module | Nalox-Comm
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23
Other Adverse Events (participants affected / at risk) | 0/25 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT04677387/Prot_SAP_002.pdf
  • Informed Consent Form (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT04677387/ICF_001.pdf